CLINICAL TRIAL: NCT03035357
Title: A Pilot Presurgical Study of Daratumumab (CD38 Antagonist) in Men With High-Risk Localized Prostate Cancer Followed by Radical Prostatectomy
Brief Title: Neoadjuvant Listeria or Daratumumab in Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI's Request
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Janssen-Cilag div. of Johnson&Johnson SE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0566
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Malignant Neoplasms of Male Genital Organs; Prostate Cancer
Keywords: Malignant neoplasms of male genital organs; Prostate cancer; Adenocarcinoma of the prostate; Daratumumab; Biomarker response
MeSH Terms: conditions — Prostatic Neoplasms | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Daratumumab (Experimental): Participants receive Daratumumab by vein over about 1 hour 1 time a week during Weeks 1-4.
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — 16 mg/kg by vein once weekly for a total of 4 doses.

SUMMARY:
The goal of this clinical research study is to learn about biomarker changes in patients who have primary prostate cancer after receiving Darzalex (daratumumab) and then have a prostatectomy (the surgical removal of the prostate) as part of their standard care. Biomarkers are found in the blood/tissue and may be related to your reaction to the study drug.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive daratumumab by vein over about 1 hour 1 time a week during Weeks 1- 4.

Length of Study:

You may receive up to 4 doses of daratumumab. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the Week 18 visit.

Study Visits:

Daratumumab treatment will interfere with blood type testing which is needed before blood transfusions can be given. For this reason, a test to find out your blood type will be performed before you receive daratumumab. You should carry the blood type card with you.

During Weeks 1 and 4:

* You will have a physical exam
* Blood (about 2 tablespoons) will be drawn for routine and blood typing.

During Weeks 2 and 3:

* You will have a physical exam.
* Blood (about 2 tablespoons) will be drawn for routine tests and for blood type testing.

During Week 6 (the week of your surgery):

* You will have a physical exam
* Blood (about 2 tablespoons) will be drawn for routine tests, including measurements of your PSA and testosterone levels. Part of this sample will also be used for blood type testing.
* You will have surgery to remove your prostate. You will sign a separate consent form explaining the procedure and its risks in more detail.

During Week 12, blood (about 2 tablespoons) will be drawn for routine tests, including measurements of your PSA and testosterone levels.

Follow-Up:

At Week 18, you will come to the clinic and asked about any side effects and how you are doing.

This is an investigational study. Daratumumab is FDA approved and commercially available to treat multiple myeloma (MM). It is considered investigational to use daratumumab in patients with prostate cancer.

The study doctor can explain how the study drug is designed to work.

Up to 15 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Consent to MD Anderson laboratory protocol PA13-0291.
2. Histological documentation of adenocarcinoma of the prostate reviewed at MD Anderson Cancer Center. Patients with small cell, neuroendocrine, or transitional cell carcinomas are not eligible.
3. Patients with high-risk prostate cancer (at least 1 core with Gleason sum >/=8) must have at least three core biopsies involved with cancer (a minimum of 6 core biopsies, must be obtained at baseline). A prostate biopsy within 3 months from screening is allowed for entry requirements.
4. No evidence of metastatic disease as documented by technetium-99m (99mTc) bone scan and by computed tomography (CT) or magnetic resonance imaging (MRI) scans.
5. Eugonadal state (serum testosterone >150 ng/dL).
6. Localized or locally advanced disease deemed by the surgeon to be resectable. Patients must be appropriate candidates for radical prostatectomy plus pelvic lymph node dissection.
7. No prior treatment for prostate cancer including prior surgery (excluding transurethral resection of the prostate [TURP]), cryoablation, pelvic lymph node dissection, radiation therapy, hormonal therapy or chemotherapy.
8. Subject must be a man age >/= 18 years of age.
9. To avoid risk of drug exposure through the ejaculate (even men with vasectomies), subjects must use a condom during sexual activity while on study drug and for 3 months following the last dose of study drug. If the subject is engaged in sexual activity with a woman of childbearing potential, a condom is required along with another effective contraceptive method consistent with local regulations regarding the use of birth control methods for subjects participating in clinical studies and their partners. Donation of sperm is not allowed while on study drug and for 3 months following the last dose of study drug.
10. ECOG performance status (PS) grade of 0 or 1.
11. Clinical laboratory values at screening: a) Hemoglobin, platelet count, absolute neutrophil count, absolute lymphocyte count within institutional normal limits. Administration of growth factors or blood transfusions will not be allowed to confirm eligibility b) Serum chemistries, renal and liver panels within institutional normal limits or requirements for radical prostatectomy
12. Each subject must sign an informed consent form (ICF) indicating that he understands the purpose of and procedures required for the study and is willing to participate in the study.

Exclusion Criteria:

1. Prior hormone therapy for prostate cancer including orchiectomy, antiandrogens, ketoconazole, or estrogens (5-alpha reductase inhibitors allowed), or LHRH agonists/antagonists.
2. Currently enrolled in another interventional study.
3. Concurrent treatment with systemic corticosteroids (prednisone dose >10 mg per day or equivalent) or other immunosuppressive drugs <14 days prior to treatment initiation. Steroids that are topical, inhaled, nasal (spray), or ophthalmic solution are permitted.
4. History of or known or suspected autoimmune disease (exception(s): subjects with vitiligo, resolved childhood atopic dermatitis, hypothyroidism, or hyperthyroidism that is clinically euthyroid at screening are allowed).
5. Known evidence of an active infection requiring systemic therapy such as human immunodeficiency virus (HIV), active hepatitis, or fungal infection.
6. History of clinically significant cardiovascular disease including, but not limited to: a) Myocardial infarction or unstable angina </= 6 months prior to treatment initiation b) Clinically significant cardiac arrhythmia c) Deep vein thrombosis, pulmonary embolism, stroke </= 6 months prior to treatment initiation d) Congestive heart failure (New York Heart Association class III-IV) e)Pericarditis/clinically significant pericardial effusion f) Myocarditis g) Endocarditis
7. History of major implant(s) or device(s), including but not limited to: a) Prosthetic heart valve(s) b) Artificial joints and prosthetics placed </= 12 months prior to treatment initiation c) Current or prior history of infection or other clinically significant adverse event associated with an exogenous implant or device that cannot be removed
8. Other prior malignancy (exceptions: adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, or any other cancer in situ currently in complete remission) </= 2 years prior to enrollment.
9. Any condition that in the opinion of the investigator, would preclude participation in this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2017-03-01 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Biomarker Response of CD3 and CD68 Following Treatment with Daratumumab. | Baseline and at 12 weeks after prostatectomy
  Biomarker response if either CD3 or CD68 has a 1.5 fold increase at prostatectomy (after treatment) compared to baseline (pre-treatment).

SECONDARY OUTCOMES:
Number of Adverse Events with Daratumumab (Adverse events as per CTCAE v4.03) | 4 weeks
  Adverse events as per CTCAE v4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Sumit K. Subudhi, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org